CLINICAL TRIAL: NCT00619346
Title: Randomized, Double-Blind Phase 1 Safety and Tolerability Study of Pafuramidine Maleate (DB289) in Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: FDA Full Clinical Hold due to safety concerns, as of 12/21/07
Sponsor: Immtech Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: C05-013
Record Dates: First submitted 2008-02-08; First posted 2008-02-20 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Healthy
Keywords: Safety; Tolerability; Assessment of potential adverse events and/or laboratory abnormalities

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Placebo tablets resembling 100 mg tablet of active drug BID X 14 days
  Interventions: Drug: Placebo
- 2 (Active Comparator): Pafuramidine maleate, 100 mg tablet, BID X 14 days
  Interventions: Drug: pafuramidine maleate

INTERVENTIONS:
Drug: Placebo — Placebo tablets, BID X 14 days
  Arms: 1
Drug: pafuramidine maleate — Pafuramidine maleate, 100 mg tablet BID X 14 days
  Arms: 2

SUMMARY:
This is a phase 1 study to establish the safety and tolerability profile of pafuramidine maleate 100 mg BID administered orally for 14 days to healthy subjects

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double-blind, placebo-controlled, parallel treatment single center safety and tolerability study. Subjects who meet all inclusion criteria and none of the exclusion criteria will be randomized in a 4:1 fashion to receive either pafuramidine maleate 100 mg tablets or matching placebo tablets administered twice daily for 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female volunteers a minimum of 18 years to 75 years of age
2. Female must be non-lactating and either be of non-child-bearing potential (i.e. sterilized via hysterectomy or bilateral tubal ligation) or if of child-bearing potential, must have a negative human chorionic gonadotropin (hCG) pregnancy test and be practicing effective dual barrier contraceptive method from consent to 42 days after initiation of study drug administration.
3. Negative test for hepatitis B surface antigen, Hepatitis C antibody and HIV 1 and 2 antibody within 14 days prior to admission to this study
4. The subject has provided written informed consent prior to admission into this study.

Exclusion Criteria:

1. History of clinically relevant medical illnesses that in the Investigator opinion may jeopardize subject safety or interfere with participation in the study, including but not limited to hemoglobinopathy, hemophilia, clinically significant retinal abnormalities, liver diseases, chronic pulmonary diseases, significant cardiovascular diseases, diabetes, thyroid diseases, gout, psychiatric or psychological disorders, CNS trauma or active seizure disorders, allergic or immunologically-mediated disorders
2. History of drug or alcohol abuse, (* 10 drinks weekly)
3. Blood donation within 30 days prior to dosing
4. History of drug allergies, anaphylaxis or laryngeal edema
5. Use of any medication within 7 days before dosing with study medication or anticipated need for any medication during the study conduct
6. Use of any investigational medication within 6 weeks prior to dosing with study medication or scheduled to receive an investigational drug other than pafuramidine maleate during the course of this study
7. Clinically significant abnormal laboratory value at screening including CBC, blood chemistry or urinalysis
8. Clinically significant anomalies noted on physical examination or ECG
9. Resting pulse rate of > 100 beats per minute or < 45 beats per minute during the screening period, either supine or standing.
10. Any condition, which compromises ability to give informed consent or to communicate with the Investigator as required for the completion of this study
11. The subject has been previously enrolled in this study. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to establish the safety and tolerability profile of pafuramidine maleate 100 mg BID administered orally for 14 days to healthy subjects. | Day 1 - Day 42

SECONDARY OUTCOMES:
The secondary objective of this study is to evaluate the potential effect of pafuramidine maleate on specific analytes that can be assessed by clinical chemistry and hematology testing. | Screening, Day 7, Day 14, Day 21 and Day 42 of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Anina M Van der Bijil, MD, Principal Investigator — Farmovs-Parexel Clinical Research Organization
Locations (1):
- Farmovs-Parexel, Bloemfontein, Republic of South Africa, South Africa